CLINICAL TRIAL: NCT01210274
Title: Characterization of the Mechanisms of Action of Resistance to Azacitidine in High-risk Myelodysplastic Syndromes and Acute Myeloid Leukemia With Multilineage Dysplasia
Brief Title: Characterization of the Mechanisms of Resistance to Azacitidine
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 10-PP-10
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Myelodysplastic Syndromes or Acute Myeloid Leukemia With Multilineage Dysplasia
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bone marrow samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Myelodysplastic syndromes (MDS) are frequent diseases in elderly patients (median age: 71 years). IPSS classification defines low risk (Low and Intermediate 1), and high risk (Intermediate 2 and High) MDS. High-risk MDS (MDS-HR) have a high risk of transformation into acute leukemia with multilineage dysplasia (AML-DML). The success of Azacitidine has been mainly achieved through a rigorous empirical and clinical research, but the molecular mechanisms by which this molecule exerts its effects remain poorly characterized. The primary mode of action of Azacytidine is through DNA demethylation, and integration in to mRNA that favor traduction inhibition. The impact of this molecule on various cell death programs involved in the elimination of leukemic cells : apoptosis and autophagy is currently poorly known.

The research program and clinical studies we proposed focus on two major aspects:

- Main objective: Molecular mechanism of action and resistance to Azacitidine: Role of apoptosis versus autophagy.

- Secondary Objective: Reversion of Azacytidine resistance using different drugs targeting apoptosis and/or autophagy. Our laboratory has identified new molecules to selectively induce different types of cell death (apoptosis or autophagy).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* High Risk or Intermediate 2 MDS (IPSS)
* AML-MD (WHO classification)
* Treatment with minimum three to six cycles of Azacitidine
* Informed consent form signed

Exclusion Criteria:

* Treatment with others chemotherapies alone or in association

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myelodysplastic syndromes or acute myeloid leukemia with multilineage dysplasia treated with Azacitidine
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
hematological response | at 3 months
  Hematological response evaluated by the International Working Group (IWG) response of Cheson
hematological response | at 6 months
  Hematological response evaluated by the International Working Group (IWG) response of Cheson

SECONDARY OUTCOMES:
Overall survival | Day 1 of treatment
  Overall survival (OS) defined as the time from start of treatment
Overall survival | at the death
  Overall survival (OS) defined as the time from start of treatment

CONTACTS AND LOCATIONS:
Locations (4):
- France (3):
  - CH d'Antibes, Antibes
  - CHU de Nice - Hôpital de l'Archet, Nice
  - Centre Antoine Lacassagne, Nice
- CH Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cluzeau T, Robert G, Mounier N, Karsenti JM, Dufies M, Puissant A, Jacquel A, Renneville A, Preudhomme C, Cassuto JP, Raynaud S, Luciano F, Auberger P. BCL2L10 is a predictive factor for resistance to azacitidine in MDS and AML patients. Oncotarget. 2012 Apr;3(4):490-501. doi: 10.18632/oncotarget.481. PMID 22577154